CLINICAL TRIAL: NCT01464697
Title: Oral Micronized Progesterone for Perimenopausal Vasomotor Symptoms
Brief Title: Progesterone for Perimenopausal Night Sweats
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Jerilynn Prior, Principal Investigator, University of British Columbia
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H10-02975
Record Dates: First submitted 2011-10-31; First posted 2011-11-03 (Estimated); Results first posted 2019-12-16 (Actual); Last update posted 2019-12-16 (Actual); Status verified 2019-11

CONDITIONS: Hot Flushes; Night Sweats
Keywords: hot flushes/hot flashes; night sweats; sleep problems; negative mood; anxiety; perimenopause; progesterone; vasomotor symptoms; depression; women's perceived change; perimenopause interference questionnaire
MeSH Terms: conditions — Hot Flashes; Parasomnias; Anxiety Disorders; Depression | interventions — Progesterone; Utrogestan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- oral micronized progesterone (Experimental): Oral micronized progesterone is Prometrium 300 mg at bedtime daily
  Interventions: Drug: Oral micronized progesterone
- Placebo Comparator (Placebo Comparator): Placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Oral micronized progesterone — 300 mg as 3-100 mg capsules taken orally at bedtime daily for 12 weeks
  Other Names: Prometrium; Utrogestan
  Arms: oral micronized progesterone
Drug: placebo — placebo comparator, taken as 3 round capsules at bedtime daily for 12 weeks
  Arms: Placebo Comparator

SUMMARY:
The purpose of this study is to test whether a oral micronized progesterone reduces the Vasomotor Symptom Score comprised of the number and severity of hot flushes and night sweats in perimenopausal women. Oral micronized progesterone is molecularly identical to human progesterone, a steroid hormone. It is sold by prescription for use to prevent endometrial cancer in women taking estrogen in menopause. This research study will test whether progesterone reduces perimenopausal hot flushes and night sweats. It will also test whether progesterone improves sleep disturbances and anxiety.

DETAILED DESCRIPTION:
This is a randomized, double-blind placebo-controlled trial of oral micronized progesterone (300 mg daily at bedtime) for perimenopausal women living anywhere in Canada. Using the self-reported maximum menstrual cycle length in the previous year, women will be stratified as in Early Perimenopause (<60 days) or Late Perimenopause (>=60 days). The design includes a 28-day baseline run-in followed by 12 weeks of randomized therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Between 35-58 years of age
2. At least 4 vasomotor symptoms (VMS) per day, on average, for at least 2/4 weeks or at least 56 over a four-week period. In addition, women should report having VMS of moderate or severe rather than mild intensity. Women reporting fewer VMS than this, but who report night sweats that awaken them from sleep on two or more nights per week will also be included.
3. Perimenopausal status either based on irregularity of menstrual periods, or by onset of new perimenopausal symptoms in women with regular periods.
4. At least one menstrual period within 12 months of study enrollment
5. Ability and willingness to complete the Daily Perimenopause Hot Flush Calendar recording instrument.
6. Ability to understand, speak, read and write English.
7. Women who are at high risk for breast cancer (ie first degree relative with breast cancer, known/suspected history of breast cancer) will be required to have a normal mammogram and clinical breast examination within 12 months of study enrollment.

Exclusion Criteria:

1. VMS without perimenopausal etiology.
2. Women who have had a hysterectomy and/or ovariectomy.
3. Peanut allergy (because peanut oil is used in the progesterone formulation.)
4. Current or recent (within the last 6-mos.) use of hormonal therapies (estrogen, progesterone, hormonal contraceptives, hormonal fertility treatments), or plans to initiate use during the study period. Two exceptions: women using progestin-releasing intrauterine device (IUD) will not be excluded as it is felt that level of hormone released will not have an effect on VMS and women taking very low-dose transdermal progesterone therapies who have VMS and meet inclusion criteria will be considered on a case-by-case basis. If enrolled, women with these exclusion exceptions will be required to continue and document use of these therapies throughout the entire trial.
5. Planned pregnancy or fertility treatment during the study period.
6. Women who are breastfeeding.
7. Participants with a score greater or equal to 15 on the Personal Health Questionnaire (PHQ-9) will be assessed on a case-by-case basis. Women assessed as needing further investigation and/or treatment for depression will be excluded.

Ages: 35 Years to 58 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 249 (Actual)
Dates: Start 2011-10; Primary Completion 2018-06-01 (Actual); Study Completion 2018-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jerilynn C Prior, MD, FRCPC, Principal Investigator — University of British Columbia
Locations (1):
- Participation from home or in-person at University of British Columbia/Centre for Menstrual Cycle and Ovulation Research (CeMCOR)/Women's Health Research Institute, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Prior JC, Hitchcock, CL. Progesterone for Vasomotor Symptoms: A 12-week Randomized, Masked Placebo-controlled Trial in Healthy, Normal-Weight Women 1-10 Years Since Final Menstrual Flow (Abstract). Endocrine Reviews 31(3): S51, 2010.
- [Background] Hitchcock CL, Prior JC. Oral micronized progesterone for vasomotor symptoms--a placebo-controlled randomized trial in healthy postmenopausal women. Menopause. 2012 Aug;19(8):886-93. doi: 10.1097/gme.0b013e318247f07a. PMID 22453200
- [Background] Prior JC, Cameron A, Hitchcock CL, et al. Oral Micronized Progesterone Beneficial for Perimenopausal Hot Flushes/Flashes and Night Sweats. Endocrine Reviews 2018;39(2) Abstract-oral presentation at Endocrine Society Conference, Chicago, 2018.
- See also: Centre for Menstrual Cycle and Ovulation Research — http://www.cemcor.ca

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Enrollment required meeting eligibility criteria by screening questionnaire but also required eligible hot flushes and night sweats on a 28-day Calendar. The difference between the listed enrolled and those who were randomized represents this fact.
Period: Overall Study
Arm/Group | Oral Micronized Progesterone | Placebo Comparator
Started | 93 | 96
Completed | 90 | 86
Not Completed | 3 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Oral Micronized Progesterone | Placebo Comparator | Total
Number analyzed (Participants) | 93 | 96 | 189
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 93 | 96 | 189
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.4 (5.0) | 50.4 (4.2) | 49.9 (4.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 93 | 96 | 189
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 2 | 9 | 11
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 83 | 82 | 165
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 4 | 8
Region of Enrollment [Number; unit: participants]
  Canada | 93 | 96 | 189

OUTCOME MEASURES:

1. Primary Outcome: Vasomotor Symptoms (VMS)/ VMS Score - at 12 Weeks
Description: Participants will complete a daily calendar (Daily Perimenopause Hot Flush Calendar) to record frequency (actual number) and severity (quantified by ordinal scale ie 0=none to 4=extreme) of hot flushes and night sweats. The VMS Score will be calculated as follows:
  Daily VMS Score = (# night sweats) x (severity) + (#hot flushes) x (severity).
  Outcome is the average daily VMS Score during the final 28 days of therapy, to be analysed with 28-day run-in scores as covariate.
Time Frame: 12 weeks
Population: Intent to Treat Population
Measure: Mean (Standard Deviation); unit: Units of Vasomotor Symptom Score
Arm/Group | Oral Micronized Progesterone | Placebo Comparator
Number analyzed (Participants) | 93 | 96
Units of Vasomotor Symptom Score | 5.5 (8.2) | 7.1 (10.4)

2. Primary Outcome: Frequency of VMS
Description: Frequency (count) of hot flushes/hot flashes and night sweats per day from prospective daily calendar records. Outcome is the average daily VMS Frequency (day + night) during the final 28 days of therapy, to be analysed with 28-day run-in scores as covariate.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: episodes per day
Arm/Group | Oral Micronized Progesterone | Placebo Comparator
Number analyzed (Participants) | 93 | 96
episodes per day | 2.4 (2.7) | 3.0 (3.7)

3. Primary Outcome: Severity of VMS
Description: Severity (0-4, 0=no intensity, 4=extreme intensity) of hot flushes/hot flashes and night sweats per day from prospective daily calendar records. Daily summary score is the maximum of daytime and nighttime severity. Outcome is the average daily severity during the final 28 days of therapy, to be analysed with 28-day run-in scores as covariate.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: Units on a Scale of 0-4
Arm/Group | Oral Micronized Progesterone | Placebo Comparator
Number analyzed (Participants) | 93 | 96
Units on a Scale of 0-4 | 1.4 (1.0) | 1.5 (1.0)

4. Primary Outcome: VMS Score by Early Perimenopause
Description: subgroup analysis of VMS Score by Early Perimenopause (no skipped period or <60 day cycle length). Outcome is the average daily VMS Score during the final 28 days of therapy, to be analysed with 28-day run-in scores as covariate. Participants will complete a daily calendar (Daily Perimenopause Hot Flush Calendar) to record frequency (actual number) and severity (quantified by ordinal scale ie 0=none to 4=extreme) of hot flushes and night sweats. The VMS Score will be calculated as follows: Daily VMS Score = (# night sweats) x (severity) + (#hot flushes) x (severity).
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: Units of Vasomotor Symptom Score
Arm/Group | Oral Micronized Progesterone | Placebo Comparator
Number analyzed (Participants) | 29 | 34
Units of Vasomotor Symptom Score | 4.4 (7.4) | 3.9 (4.0)

5. Primary Outcome: VMS Score by Late Perimenopause
Description: subgroup analysis of VMS Score by Late Perimenopause (those with skipped or ≥60 day cycle lengths). Outcome is the average daily VMS Score during the final 28 days of therapy, to be analysed with 28-day run-in scores as covariate. Participants will complete a daily calendar (Daily Perimenopause Hot Flush Calendar) to record frequency (actual number) and severity (quantified by ordinal scale ie 0=none to 4=extreme) of hot flushes and night sweats. The VMS Score will be calculated as follows: Daily VMS Score = (# night sweats) x (severity) + (#hot flushes) x (severity).
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: Units of Vasomotor Symptom Score
Arm/Group | Oral Micronized Progesterone | Placebo Comparator
Number analyzed (Participants) | 64 | 62
Units of Vasomotor Symptom Score | 5.9 (8.5) | 8.8 (12.3)

6. Primary Outcome: Subgroup Analysis for Those With Frequent and Severe VMS - VMS Score
Description: VMS Score for those with more frequent (≥7 per day and moderate to severe episodes of intensity 2-4) at baseline. Participants will complete a daily calendar (Daily Perimenopause Hot Flush Calendar) to record frequency (actual number) and severity (quantified by ordinal scale ie 0=none to 4=extreme) of hot flushes and night sweats. The VMS Score will be calculated as follows:
  Daily VMS Score = (# night sweats) x (severity) + (#hot flushes) x (severity).
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: Units of Vasomotor Symptom Score
Arm/Group | Oral Micronized Progesterone | Placebo Comparator
Number analyzed (Participants) | 19 | 16
Units of Vasomotor Symptom Score | 11.8 (9.0) | 15.1 (17.1)

7. Secondary Outcome: Sleep Problems
Description: Daily average rating of sleep problems (0-4) from prospective daily calendar records.
  Outcome is the average daily rating during the final 28 days of therapy, to be analysed with 28-day run-in scores as covariate. Scale name: Sleep Problems (4=Worst, 0=None)
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: Units on a ordinal Scale
Arm/Group | Oral Micronized Progesterone | Placebo Comparator
Number analyzed (Participants) | 93 | 96
Units on a ordinal Scale | 0.8 (0.8) | 1.0 (0.9)

8. Secondary Outcome: Anxiety
Description: Daily average rating of anxiety (0-4) from prospective daily calendar records. Outcome is the average daily rating during the final 28 days of therapy, to be analysed with 28-day run-in scores as covariate. Scale name: Anxiety (4=Worst, 0=None)
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: Units on a ordinal Scale
Arm/Group | Oral Micronized Progesterone | Placebo Comparator
Number analyzed (Participants) | 93 | 96
Units on a ordinal Scale | 0.5 (0.6) | 0.6 (0.8)

9. Secondary Outcome: Women's Perceived Changes in Daytime Hot Flushes for Whole Population
Description: Women's Perceived Changes Questionnaire of changes (from -5 to 0 to +5) in Daytime Hot Flushes (both number and severity) as recorded on the Final Questionnaire.
  Scale Name: Daytime Hot Flush Change Decrease is -5 to -1; No change is 0; Increase is +1 to +5. This is women's perception of the change from run-in to when they recorded it at the end of the trial (at 12 weeks).
  No calculation is needed.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: Change Scale -5 to +5, no change is 0
Arm/Group | Oral Micronized Progesterone | Placebo Comparator
Number analyzed (Participants) | 90 | 86
Change Scale -5 to +5, no change is 0 | -2.3 (2.3) | -1.8 (2.3)

10. Secondary Outcome: Women's Perceived Changes in Night Sweats for Whole Population
Description: Women's Perceived Changes Questionnaire of changes (from -5 to 0 to +5) in Nighttime Night Sweats (both number and severity) as recorded on the Final Questionnaire.
  Scale Name: Night Sweats Change Decrease is -5 to -1; No change is 0; Increase is +1 to +5. This is women's perception of the change from run-in to when they recorded it at the end of the trial (at 12 weeks).
  No calculation is needed.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: Change Scale -5 to +5, no change is 0
Arm/Group | Oral Micronized Progesterone | Placebo Comparator
Number analyzed (Participants) | 90 | 86
Change Scale -5 to +5, no change is 0 | -2.5 (2.0) | -1.9 (2.0)

11. Secondary Outcome: Women's Perceived Changes in Quality of Sleep for Whole Population
Description: Women's Perceived Changes Questionnaire of changes (from -5 to 0 to +5) in the quality of sleep over the three months of the trial as assessed by the Final Questionnaire based on their random assignment to the progesterone or placebo arms of this RCT (Randomized Controlled Trial) and by Early/Late perimenopause.
  Scale Name: Quality of Sleep Change Decrease is -5 to -1; No change is 0; Increase is +1 to +5. This is women's perception of the change from run-in to when they recorded it at the end of the trial (at 12 weeks).
  No calculation is needed.
Time Frame: 12 weeks
Measure: Mean (Full Range); unit: Change Scale -5 to +5, no change is 0
Arm/Group | Oral Micronized Progesterone | Placebo Comparator
Number analyzed (Participants) | 90 | 86
Change Scale -5 to +5, no change is 0 | 2.0 [0.0 to 4.0] | 0.0 [0.0 to 3.0]

12. Secondary Outcome: Perception of Interference of Overall Perimenopausal Changes With Usual Activities in Women
Description: Final perceptions of interference of overall perimenopausal changes with usual activities (as recorded by the CeMCOR PIQ - Centre for Menstrual Cycle and Ovulation Research Perimenopause Interference Questionnaire) at 12 weeks in women randomized to the progesterone versus to placebo.
  Scale Name: Perceived Interference Score: 100 mm line (0 = No Interference; 100 = Severe Interference)
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: Visual Analogue scale 0-100 mm
Arm/Group | Oral Micronized Progesterone | Placebo Comparator
Number analyzed (Participants) | 93 | 96
Visual Analogue scale 0-100 mm | 22.6 (18.3) | 28.2 (21.7)

13. Secondary Outcome: Perception of Interference of Overall Perimenopausal Changes With Usual Activities in Women - Early Perimenopause
Description: Final perceptions of interference of overall perimenopausal changes with usual activities (as recorded by the CeMCOR Perimenopause Interference Questionnaire [CeMCOR PIQ]) at 12 weeks in women randomized to the progesterone versus to placebo.
  Scale Name: Perceived Interference Score: 100 mm line (0 = No Interference; 100 = Severe Interference)
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: Visual Analogue scale 0-100 mm
Arm/Group | Oral Micronized Progesterone | Placebo Comparator
Number analyzed (Participants) | 29 | 34
Visual Analogue scale 0-100 mm | 25.7 (20.2) | 33.0 (22.7)

14. Secondary Outcome: Perception of Interference of Overall Perimenopausal Changes With Usual Activities in Women - Late Perimenopause
Description: as for outcome 13
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: Visual Analogue scale 0-100 mm
Arm/Group | Oral Micronized Progesterone | Placebo Comparator
Number analyzed (Participants) | 64 | 62
Visual Analogue scale 0-100 mm | 21.3 (17.5) | 25.6 (20.9)

15. Secondary Outcome: Perception of Interference of Perimenopausal Body Changes With Usual Activities in Women
Description: Final perceptions of interference of perimenopausal body changes with usual activities (as recorded by the CeMCOR Perimenopause Interference Questionnaire [CeMCOR PIQ]) in women randomized to the progesterone versus to placebo.
  Scale Name: Perceived Interference Score: 100 mm line (0 = No Interference; 100 = Severe Interference)
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: Visual Analogue scale 0-100 mm
Arm/Group | Oral Micronized Progesterone | Placebo Comparator
Number analyzed (Participants) | 93 | 96
Visual Analogue scale 0-100 mm | 22.4 (20.1) | 27.8 (24.2)

16. Secondary Outcome: Perception of Interference of Perimenopausal Mood Changes With Usual Activities in Women
Description: Final perceptions of interference of perimenopausal mood changes with usual activities (as recorded by the CeMCOR Perimenopause Interference Questionnaire [CeMCOR PIQ]) in women randomized to the progesterone versus to placebo.
  Scale Name: Perceived Interference Score: 100 mm line (0 = No Interference; 100 = Severe Interference)
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: Visual Analogue scale 0-100 mm
Arm/Group | Oral Micronized Progesterone | Placebo Comparator
Number analyzed (Participants) | 93 | 96
Visual Analogue scale 0-100 mm | 22.7 (20.1) | 29.3 (23.5)

17. Secondary Outcome: Women's Perceived Changes in Daytime Hot Flushes in Early Perimenopause
Description: Women's Perceived Changes Questionnaire of changes (from -5 to 0 to +5) in Daytime Hot Flushes (both number and severity) as recorded on the Final Questionnaire and by subgroup for Early Perimenopause.
  Scale Name: Perceived Daytime Hot Flush Change Decrease is -5 to -1; No change is 0; Increase is +1 to +5.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: Change Scale -5 to +5, no change is 0
Arm/Group | Oral Micronized Progesterone | Placebo Comparator
Number analyzed (Participants) | 26 | 30
Change Scale -5 to +5, no change is 0 | -1.7 (2.9) | -1.3 (1.8)

18. Secondary Outcome: Women's Perceived Changes in Night Sweats in Early Perimenopause
Description: Women's Perceived Changes Questionnaire of changes (from -5 to 0 to +5) in Nighttime Night Sweats (both number and severity) as recorded on the Final Questionnaire and by subgroup for Early Perimenopause.
  Scale Name: Perceived Night Sweats Change Decrease is -5 to -1; No change is 0; Increase is +1 to +5.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: Change Scale -5 to +5, no change is 0
Arm/Group | Oral Micronized Progesterone | Placebo Comparator
Number analyzed (Participants) | 26 | 30
Change Scale -5 to +5, no change is 0 | -2.9 (1.9) | -1.9 (1.6)

19. Secondary Outcome: Women's Perceived Changes in Daytime Hot Flushes in Late Perimenopause
Description: Women's Perceived Changes Questionnaire of changes (from -5 to 0 to +5) in Daytime Hot Flushes (both number and severity) as recorded on the Final Questionnaire and by subgroup for Late Perimenopause.
  Scale Name: Perceived Daytime Hot Flush Change Decrease is -5 to -1; No change is 0; Increase is +1 to +5.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: Change Scale -5 to +5, no change is 0
Arm/Group | Oral Micronized Progesterone | Placebo Comparator
Number analyzed (Participants) | 64 | 56
Change Scale -5 to +5, no change is 0 | -2.5 (2.1) | -2.0 (2.4)

20. Secondary Outcome: Women's Perceived Changes in Night Sweats in Late Perimenopause
Description: Women's Perceived Changes Questionnaire of changes (from -5 to 0 to +5) in Nighttime Night Sweats (both number and severity) as recorded on the Final Questionnaire and by subgroup for Late Perimenopause.
  Scale Name: Perceived Night Sweats Change Decrease is -5 to -1; No change is 0; Increase is +1 to +5.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: Change Scale -5 to +5, no change is 0
Arm/Group | Oral Micronized Progesterone | Placebo Comparator
Number analyzed (Participants) | 64 | 56
Change Scale -5 to +5, no change is 0 | -2.4 (2.1) | -1.9 (2.2)

21. Secondary Outcome: Depression Related to Progesterone Therapy in Whole Population
Description: Final PHQ9 (Personal Health Questionnaire 9) Score for Depression related to progesterone therapy in perimenopause will be assessed based on the Personal Health Questionnaire-9 (PHQ-9) score changes within-woman from baseline to the end-of-trial on progesterone compared with placebo.
  Scale Name: PHQ9 Scale (0 = No Depression; 27 = Severe Depression)
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: PHQ9 Scale: 0-27
Arm/Group | Oral Micronized Progesterone | Placebo Comparator
Number analyzed (Participants) | 93 | 96
PHQ9 Scale: 0-27 | 4.8 (4.4) | 5.4 (4.3)

22. Secondary Outcome: Depression Related to Progesterone Therapy in Early Perimenopause
Description: Final PHQ9 Score for Depression related to progesterone therapy in Early Perimenopause will be assessed based on the Personal Health Questionnaire-9 (PHQ-9) score changes within-woman from baseline to the end-of-trial on progesterone compared with placebo.
  Scale Name: PHQ9 Scale (0 = No Depression; 27 = Severe Depression)
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: PHQ9 Scale: 0-27
Arm/Group | Oral Micronized Progesterone | Placebo Comparator
Number analyzed (Participants) | 29 | 34
PHQ9 Scale: 0-27 | 6.0 (4.6) | 5.4 (3.6)

23. Secondary Outcome: Depression Related to Progesterone Therapy in Late Perimenopause
Description: Final PHQ9 Score for Depression related to progesterone therapy in Late Perimenopause will be assessed based on the Personal Health Questionnaire-9 (PHQ-9) score changes within-woman from baseline to the end-of-trial on progesterone compared with placebo.
  Scale Name: PHQ9 Scale (0 = No Depression; 27 = Severe Depression)
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: PHQ9 Scale: 0-27
Arm/Group | Oral Micronized Progesterone | Placebo Comparator
Number analyzed (Participants) | 64 | 62
PHQ9 Scale: 0-27 | 4.4 (4.3) | 5.4 (4.6)

24. Secondary Outcome: Percentage of Women With Perceived Changes in Menstrual Flow
Description: Menstrual flow related to progesterone therapy in perimenopause was assessed based on Women's Perceived Changes Questionnaire of changes in the experience of menstrual flow/vaginal bleeding from the Final Questionnaire.
Time Frame: 12 weeks
Population: The discrepancy in the Number of Participants analyzed is due to missing data on the Final Questionnaire.
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Micronized Progesterone | Placebo Comparator
Number analyzed (Participants) | 90 | 86
Participants | 65 | 74

ADVERSE EVENTS:
Time Frame: From randomization until the final questionnaire the day after the last experimental therapy, up to 12 weeks.
Description: We followed Best Clinical Practice Guidelines. All reported events were included. They were blindly classified by intensity and by potential relationship with the experimental therapy.
Arm/Group | Oral Micronized Progesterone | Placebo Comparator
All-Cause Mortality (participants affected / at risk) | 0/93 | 0/96
Serious Adverse Events (participants affected / at risk) | 0/93 | 0/96
Other Adverse Events (participants affected / at risk) | 22/93 | 8/96
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Oral Micronized Progesterone (N=93) | Placebo Comparator (N=96)
Musculoskeletal, arthritis, connective tissue issues (Musculoskeletal and connective tissue disorders) | 6 | 1
Nausea, GI tract problems (Gastrointestinal disorders) | 8 | 1
Dizziness (General disorders) | 1 | 1
Edema, atrial fibrillation, increased blood pressure, and headache (Cardiac disorders) | 5 | 3
Worsening VMS (Reproductive system and breast disorders) | 0 | 1
Post-traumatic stress (Psychiatric disorders) | 0 | 1
Probable depression (Psychiatric disorders) | 1 | 0
Facial acne (Skin and subcutaneous tissue disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
Given no previous RCT of VMS only in perimenopause, despite a blinded study assessment, we were still under powered. Women's Perceived Changes assessments, were not congruent with the VMS Score.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-18): https://cdn.clinicaltrials.gov/large-docs/97/NCT01464697/Prot_SAP_000.pdf